CLINICAL TRIAL: NCT00946244
Title: A Longitudinal Study of Effectiveness of Early Intervention for Preterm Infants
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200812114R
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2009-11

CONDITIONS: Premature Birth
Keywords: Early intervention; Mother-child interaction; Neurodevelopment; Parenting; Prematurity; Preschool age
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Term infants: Healthy term infants
- Usual care program: VLBW preterm infants who received usual medical care during hospitalization after birth
- Clinic-based intervention program: VLBW preterm infants who received specific early intervention program delivered at clinic before 1 year of corrected age (in previous study)
- Home-based intervention program: VLBW preterm infants who received specific early intervention program delivered at home before 1 year of corrected age (in previous study)

SUMMARY:
The main purpose of this study is to extend the investigators' previous research to longitudinally examine the effectiveness of three early intervention programs: usual care program, clinic-based intervention program and home-based intervention program for very low birth weight preterm children at 3 and 4 years of age. Normal weight full-term children will also be included to serve as the reference group. Effectiveness assessments will include child, parenting, and transactions measures. Child outcome measures will include health status, growth, neurodevelopment and behavior; parenting outcome measures will include parental stress, competence, efficacy and family support; transactions outcome measure will include parent-child interaction procedures.

DETAILED DESCRIPTION:
Accumulating data on early intervention for preterm infants illustrated short-term benefits on enhancing child development and decreasing parental stress, particularly for those of heavier birth weights. However, rare studies had designed early intervention program for small preterm infants and longitudinally examined the effectiveness in various outcome domains. Our research team recently conducted a clinical randomization trial on the effectiveness of three early intervention programs: usual care program (UCP), clinic-based intervention program (CBIP) and home-based intervention program (HBIP) on very low birth weight (VLBW, birth weight <1,500 g) preterm infants from the neonatal period to two years corrected age (CA). The latter two were comprehensive, intensive intervention programs that combined child- and parent-focused services beginning in hospitalization and ending at one year CA as delivered at clinic and home respectively. This three-year research project has extended our previous work to longitudinally examine the effectiveness of the three intervention programs in 180 VLBW preterm infants at 3 and 4 years of age. Sixty full-term infants will also be included to serve as the reference group. Outcome measures will include child (i.e., health, growth, neurodevelopment and behavior), parenting (i.e., parental stress, competency, efficacy and family support) and mother-child transactions (i.e., free-play and frustrating episode). The longitudinal data on the effectiveness of these early intervention programs for VLBW preterm infants will provide important information to help early intervention professionals and public policy makers to develop effective intervention for preterm children at risk for developmental problems.

ELIGIBILITY:
Inclusion Criteria:

* Body weight below 1501 gm
* Gestational age under 37 weeks
* Admission to the study hospitals within the first 7 days of life
* Singleton or the first child of twin or multiple births
* Physiologically stable at PCA 36 weeks as determined by attending physician
* Hospital discharge prior to PCA 44 weeks

Exclusion Criteria:

* Seizure
* Hydrocephalus
* Ventriculoperitoneal shunt
* Meningitis, periventricular leukomalacia
* Grade III to IV intraventricular hemorrhage
* Stage IV retinopathy of prematurity)
* Necrotizing enterocolitis with colostomy
* Severe cardiopulmonary disease requiring daily oxygen use at hospital discharge

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term and VLBW preterm children were born at the National Taiwan University Hospital and the Mackay Memorial Hospital (MMH)
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Child's development (health, growth, neurodevelopment and behavior) | 3 and 4 years of age

SECONDARY OUTCOMES:
Parenting function (parent stress, competency, efficacy and family support) | 3 and 4 years of age
Parent-child transactions | 3 and 4 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Fang Jeng, Sc.D, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Li SJ, Tsao PN, Tu YK, Hsieh WS, Yao NJ, Wu YT, Jeng SF. Cognitive and motor development in preterm children from 6 to 36 months of age: Trajectories, risk factors and predictability. Early Hum Dev. 2022 Sep;172:105634. doi: 10.1016/j.earlhumdev.2022.105634. Epub 2022 Jul 28. PMID 35921693